CLINICAL TRIAL: NCT07266961
Title: The Effects of Low-Intensity Resistance Training Combined With Blood Flow Restriction Versus Moderate-Intensity Resistance Training on Cardiorespiratory Fitness in Elderly Women
Brief Title: Low-BFR vs Moderate-Intensity Resistance Training on Cardiorespiratory Fitness in Elderly Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Soetomo General Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: DrSoetomoLIRT-BFR&MIRT
Record Dates: First submitted 2025-11-25; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-10

CONDITIONS: Cardiorespiratory Fitness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LIRT-BFR group (Experimental): The LIRT-BFR group used a cuff on the upper third of the thigh with a restriction pressure of 50 mmHg or 40% Arterial Occlusion Pressure to apply BFR while engaging in low-load resistance training that targeted the quadriceps femoris muscle at an intensity of 20-30% of 1-RM. The resistance training protocol consists of four sets of knee extensions using an ankle weight in a sitting position. Each set consists of 30 repetitions on the first set and 15 repetitions each on sets 2-4 with a 30-second interval between sets. The air pressure cuff was deflated during the interval period. In the third week, the weight load was recalculated to 40% of 1-RM in order to accommodate subsequent 1-RM testing procedures.
  Interventions: Other: Low Intensity Resistance Training and Blood Flow Resistance
- MIRT group (Active Comparator): The MIRT group conducted three sessions of moderate-intensity resistance training, concentrating on the quadriceps femoris muscle, with weights set at 40-60% of their 1RM or higher. While the MIRT protocol resembled that of LIRT-BFR, each session comprised 8-12 repetitions, followed by a 2-minute rest between sets. In the third week, the 1-RM testing protocol was revised, with the weight adjusted to 60% of the 1-RM.
  Interventions: Other: Moderate Intensity Resistance Training

INTERVENTIONS:
Other: Low Intensity Resistance Training and Blood Flow Resistance — The LIRT-BFR group used a cuff on the upper third of the thigh with a restriction pressure of 50 mmHg or 40% Arterial Occlusion Pressure to apply BFR while engaging in low-load resistance training that targeted the quadriceps femoris muscle at an intensity of 20-30% of 1-RM. The resistance training protocol consists of four sets of knee extensions using an ankle weight in a sitting position. Each set consists of 30 repetitions on the first set and 15 repetitions each on sets 2-4 with a 30-second interval between sets. The air pressure cuff was deflated during the interval period. In the third week, the weight load was recalculated to 40% of 1-RM in order to accommodate subsequent 1-RM testing procedures.
  Arms: LIRT-BFR group
Other: Moderate Intensity Resistance Training — The MIRT group conducted three sets of moderate-intensity resistance training, concentrating on the quadriceps femoris muscle, with weights set at 40-60% of their 1RM or higher. While the MIRT protocol resembled that of LIRT-BFR, each set comprised 8-12 repetitions, followed by a 2-minute rest between sets. In the third week, the 1-RM testing protocol was revised, with the weight adjusted to 60% of the 1-RM.
  Arms: MIRT group

SUMMARY:
This study is aiming to compare the CRF utilizing LIRT-BFR and MIRT in the elderly. Both techniques provided comparable gains in VO₂ max and the BORG scale. The BFR group displayed a greater level of safety for elderly to undertake resistance training with the same benefit as the MIRT group.

DETAILED DESCRIPTION:
Decreased cardiorespiratory fitness (CRF) is a common issue among older adults and contributes to reduced physical activity levels and quality of life. While aerobic exercise is known to improve CRF, it has limited effects on muscle strength and mass. In contrast, resistance training can enhance both cardiorespiratory and muscular fitness when performed at moderate intensity. Blood flow restriction (BFR) applied during low-intensity resistance training (LIRT-BFR) has emerged as a promising alternative that may elicit similar physiological benefits to traditional moderate-intensity resistance training (MIRT) while reducing mechanical stress on joints and muscles. This study aims to compare the effects of six weeks of LIRT-BFR versus MIRT on cardiorespiratory fitness in elderly women. Twenty-eight participants were randomly assigned to either the LIRT-BFR group or the MIRT group and completed 12 supervised exercise sessions over six weeks. The MIRT group performed exercises at 40-60% of one-repetition maximum (1-RM), while the LIRT-BFR group exercised at 20-30% of 1-RM under blood flow restriction. The primary outcome was the predicted VO₂max obtained from the 6-Minute Walking Test (6MWT). The secondary outcome was the rating of perceived exertion (RPE) measured using the modified Borg scale following the 6MWT.

ELIGIBILITY:
Inclusion Criteria:

* Female aged ≥60 years who routinely performed aerobic exercise in RSUD Dr. Soetomo
* Normal cognitive function (MoCA-Ina score ≥ 26)
* Passed the screening questionnaire.

Exclusion Criteria:

* Severe physical disability (presented with a musculoskeletal, cardiorespiratory, or neurological disease that affected physical performance during exercise)
* Visual and hearing impairment
* Balance impairment
* Blood clotting disorder
* Peripheral arterial disease on the legs
* Deep vein thrombosis
* Neuropathy in the lower extremity
* Uncontrolled hypertension or diabetes mellitus
* Previous stroke and compartment syndrome
* Knee osteoarthritis with moderate pain (VAS >4)
* Past vascular surgery
* Prior skin graft on the lower leg area
* Lower limb bone surgery within the past 12 weeks
* Immobilization during the last 4 weeks
* Statin consumption
* Sarcopenia
* Benign paroxysmal positional vertigo with an exacerbation in the previous 4 weeks.

Min Age: 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
VO₂max | The VO₂max was measured before the intervention and after the intervention in the third and sixth weeks. The participants took a rest of at least 30 minutes after the resistance training to avoid fatigue in the legs, which could interfere with the 6MWD.
  The main parameter evaluated in this study is cardiorespiratory fitness using VO₂max prediction value by carrying out a 6MWT.

SECONDARY OUTCOMES:
BORG RPE Scale | RPE was measured with the BORG Scale 6-20 to determine the participant's level of difficulty and exertion after the 6 MWT. The evaluation of RPE was continued for 60 minutes as guarantee the participant's safety and to monitor the complications.
  The BORG RPE scale was used to measure a person's effort and exertion, dyspnea, and exhaustion during physical labor. RPE was measured with the BORG Scale 6-20 to determine the participant's level of difficulty and exertion after the 6 MWT.

CONTACTS AND LOCATIONS:
Overall Officials: Nuniek Nugraheni Sulistiawaty, Principal Investigator — Department of Physical Medicine and Rehabilitation - Dr. Soetomo Regional Hospital
Locations (1):
- Department of Physical Medicine and Rehabilitation - Dr. Soetomo Regional Hospital, Surabaya, East Java, Indonesia

IPD SHARING:
Plan to Share IPD: No